CLINICAL TRIAL: NCT05406453
Title: Whole Genome Sequencing of Tuberculosis for Disease Control in Madagascar - a Cluster Randomized Controlled Trial to Evaluate Different Community-wide Intervention Strategies.
Brief Title: Whole Genome Sequencing of Tuberculosis for Disease Control in Madagascar
Acronym: TB_WGS_cRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Madagascar (Other)
Collaborators: The National Tuberculosis Program, Madagascar (Unknown); Centre de Recherche du Centre Hospitalier de l'Université de Montréal (Other)
Responsible Party: Principal Investigator, Simon Grandjean Lapierre, Researcher, Institut Pasteur de Madagascar
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-01; PJT 75243 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2022-06-02; First posted 2022-06-06 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Tuberculosis
Keywords: Whole genome sequencing; cluster randomized controlled trial
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Intervention Model Description: cRCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Madagascar standard of care (No Intervention): Description :
  * Passive case finding,
  * Smear microscopy testing, and
  * household contact tracing
- Best practices (No Intervention): Description :
  * Active case finding,
  * Smear microscopy
  * Xpert MTB/RIF Ultra testing (= rapid test by Genexpert for tuberculosis (TB) and rifampin resistance (RIF-R)) and
  * household contact tracing
- Novel intervention (Experimental): Description :
  * Active case finding,
  * Smear microscopy
  * Xpert MTB/RIF Ultra testing and
  * household contact tracing
  Interventions: Other: Whole Genome Sequencing testing

INTERVENTIONS:
Other: Whole Genome Sequencing testing — Whole Genome Sequencing testing, community-based contact tracing
  Arms: Novel intervention

SUMMARY:
Tuberculosis (TB) whole genome sequencing (WGS) allows outbreak identification and disease transmission tracking.

It is hypothesized that prospective WGS-guided epidemiological investigations improve case detection compared to current best practices by adapting contact tracing strategies to local transmission patterns.

A cluster randomized controlled trial (cRCT) will be performed in high TB incidence villages of Haute Matsiatra region in Madagascar. Communities will be randomized in three separate TB control strategies comparing (1) standard of care, (2) the World Health Organization (WHO) recommended best practices and (3) a novel intervention involving TB WGS cluster-guided epidemiological investigations. The incremental value of TB WGS on case notifications and reduction of TB burden will be measured.

Secondary studies will be nested within this cRCT will include:

* A qualitative study which will increase the understanding of the factors facilitating and hindering implementation of WGS-based diagnostics within health systems.
* A cost effectiveness analysis study which will measure the cost effectiveness of newly implemented laboratory methods.

Field and genomic epidemiology data from this project will inform future work on the design of community-level TB elimination strategies in collaboration with Madagascar National TB program

ELIGIBILITY:
Inclusion Criteria:

* Subjects suspected TB
* subject living in the study area

Exclusion Criteria:

* unable to take a sputum sample

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98362 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
the total number of TB cases detected / 100 000 inhabitants | an average of 1 year
  total number of TB cases detected / 100,000 inhabitants / year in each group during the first year of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Grandjean Lapierre, MD MSc FRCPC, Principal Investigator — CHUM
Locations (1):
- Fokontany Vohibato, Vohibato, Madagascar

IPD SHARING:
Plan to Share IPD: Yes
Upon request to the investigator
Supporting Information: Study Protocol, ICF
Time Frame: Upon request
Access Criteria: Upon request to the investigator

REFERENCES:
- [Derived] Ametepe ESA, Andriamanoha N, Andrianomanana FR, Point F, Mangahasimbola RT, Dyachenko A, Hall M, Gamana TM, Knoblauch AM, Razafindrasoa YY, Nimalan A, Behr M, Durand M, Johri M, Iqbal Z, Rakotoarivelo AR, Randremanana RV, Rakotosamimanana N, Lapierre SG. Whole genome sequencing of M. tuberculosis for disease control in high-burden settings: study protocol for a cluster randomized controlled trial evaluating different community-wide intervention strategies in rural Madagascar. Trials. 2024 Oct 25;25(1):717. doi: 10.1186/s13063-024-08537-4. PMID 39456079